CLINICAL TRIAL: NCT04697134
Title: A Community-based Conscious Discipline Program to Reduce Corporal Punishment in the Caribbean
Brief Title: Community-Based Conscious Discipline Program in Grenada
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Windward Islands Research and Education Foundation (Other)
Collaborators: Grand Challenges Canada (Other); GRENCASE (Unknown); St. George's University (Unknown)
Responsible Party: Principal Investigator, Dr. Randall Waechter, Associate Director of Research, Windward Islands Research and Education Foundation
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: SGUSavingBrainsI
Record Dates: First submitted 2021-01-04; First posted 2021-01-06 (Actual); Last update posted 2021-01-07 (Actual); Status verified 2021-01

CONDITIONS: Behavior, Child; Neurocognition, Child; Development, Child
MeSH Terms: conditions — Child Behavior

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Conscious Discipline Intervention Group (Experimental): Participants in this group received one-on-one Conscious Discipline classes with a Roving Caregiver. These classes consisted of the dissemination of Conscious Discipline Skills and fun songs, games, and activities to foster connections between the infant and caregiver. Both the infant and caregiver received the intervention simultaneously.
  Interventions: Behavioral: Conscious Discipline-Based Environmental Enrichment Intervention
- Control (No Intervention): Participants in this group did not receive the intervention.

INTERVENTIONS:
Behavioral: Conscious Discipline-Based Environmental Enrichment Intervention — Conscious Discipline, a social-emotional skills-based learning program that draws on current brain research and fosters enhanced connections between parents and their children.
  Arms: Conscious Discipline Intervention Group

SUMMARY:
To improve neurocognitive outcomes in 2-year-old children by implementing a community-based intervention program that follows the principles of Conscious Discipline.

DETAILED DESCRIPTION:
We aimed to introduce Conscious Discipline (CD) in Grenada as a means of improving neurodevelopment in 2-year-old children. The CD intervention promotes improved social-emotional connections between parents/guardians and children that reduces harsh discipline and corporal punishment and provides an ideal environment for the development of higher cognitive functioning (e.g. working memory, inhibition, emotional regulation).

The intervention is implemented by using a distributed local, train-the-trainer model in partnership with the Grenada Roving Caregiver Program, managed by GRENCASE. CD training was provided to 85 existing Roving Caregivers, 70 of whom were certified as Conscious Discipline Paraprofessionals (CDPPs). Certified CDPPs traveled out to communities and villages throughout Grenada, to impart knowledge and skills to new and expecting parents.

Following the intervention, parents who received CD training were assessed in their ability to implement CD skills with their child(ren). Neurocognition was assessed in children post-intervention using the INTERGROWTH 21st Neurodevelopmental Assessment (INTERNDA). Neurocognitive outcomes were compared between the intervention arm and the waitlist control arm of the study.

ELIGIBILITY:
Inclusion Criteria:

* Participants actively enrolled in the Roving Caregiver Program (0-2-year-olds living with parents in at-risk communities served by the RCP)

Exclusion Criteria:

* Not enrolled in the Roving Caregiver Program

Ages: 22 Months to 30 Months | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 333 (Actual)
Dates: Start 2015-02-02 (Actual); Primary Completion 2016-08-18 (Actual); Study Completion 2016-08-18 (Actual)

PRIMARY OUTCOMES:
INTERGROWTH 21st Neurodevelopment Assessment (INTER-NDA) | 22-30 Months
  The INTER-NDA is a measure of cognition, motor skills (fine and gross motor), language (expressive and receptive), behavior, executive function, attention and social-emotional reactivity for 2-year-olds. The measure is comprised of 30 items scored across a spectrum, with higher scores indicating better outcomes.

CONTACTS AND LOCATIONS:
Overall Officials: Randall Waechter, PhD, Principal Investigator — Windard Islands Research and Education Foundation
Locations (1):
- Windward Islands Research and Education Foundation, Saint George's, Grenada

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Waechter R, Evans R, Fernandes M, Bailey B, Holmes S, Murray T, Isaac R, Punch B, Cudjoe N, Orlando L, Landon B. A Community-based Responsive Caregiving Program Improves Neurodevelopment in Two-year Old Children in a Middle-Income Country, Grenada, West Indies. Psychosoc Interv. 2022 May 13;31(2):97-107. doi: 10.5093/pi2022a6. eCollection 2022 May. PMID 37360060